CLINICAL TRIAL: NCT04689347
Title: Phase 1b/2 Trial of 5-fluorouracil, Leucovorin, Irinotecan in Combination With Temozolomide (FLIRT) and Bevacizumab for the First-line Treatment of Patients With MGMT Silenced, Microsatellite Stable Metastatic Colorectal Cancer.
Brief Title: 5FU/LV, Irinotecan, Temozolomide and Bevacizumab for MGMT Silenced, Microsatellite Stable Metastatic Colorectal Cancer.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INT 151/20
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Temozolomide; MGMT; microsatellite stable; First-line; Phase 1; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Leucovorin; Fluorouracil; Temozolomide

STUDY DESIGN:
Intervention Model Description: A 3 + 3 design will be used to assess the maximum tolerated dose (MTD) or maximum tested dose of the combination FLIRT-bevacizumab. The MTD will be defined as the dose level at which ≥2/3 or ≥2/6 subjects experience a dose-limiting toxicity (DLT). When the MTD or maximum tested dose has been determined or reached, the RP2D to be tested in a future phase II trial will be one dose level below the MTD or the maximum tested dose if MTD will not be reached. At least 6 patients should be treated at the RD during the dose escalation.
  Regarding the expansion part of the study, considering a 9-month PFS rate of 35% in patients receiving FOLFIRI plus bevacizumab (which has been shown in the RAS mutated subgroup of TRIBE trial and considering that MGMT methylation is strongly associated with RAS mutations), an overall sample size of 27 patients achieves an 80% power to detect the probability to increase 9-month PFS rate to 55% with a one-sided α level of 0.1 by the combination of temozolomide at
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLIRT-bevacizumab (Experimental): Bevacizumab intravenous infusion (IV), irinotecan IV, leucovorin (LV) IV, 48-hours continuous intravenous infusion of 5-fluorouracil (5-FU), given every 14 days, in combination with oral (PO) temozolomide with progressive dose escalation at inter-patient level over days 1-5 every 28 days.
  The treatment will consist of an induction period of four 28-day cycles of FLIRT- bevacizumab followed by maintenance regimen of 5-FU/LV-bevacizumab administered every 14 days in combination with PO temozolomide according to dose level over days 1-5 every 28 days in patients without progressive disease at the end of the induction period.
  In the phase 2 patient will receive the same treatment of the phase 1b with temozolomide at the RP2D (150 mg/sqm)
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5Fluorouracil; Drug: Temozolomide

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 5 mg/kg intravenous infusion every 2 weeks
Drug: Irinotecan — irinotecan 165 mg/sqm intravenous infusion every 2 weeks
Drug: Leucovorin — leucovorin 200 mg/sqm intravenous infusion every 2 weeks
Drug: 5Fluorouracil — 48-hours continuous intravenous infusion of 5-fluorouracil (5-FU) 3200 mg/sqm every 2 weeks
Drug: Temozolomide — Oral temozolomide with progressive dose escalation at inter-patient level over days 1-5 every 28 days. (75 mg/sqm; 100 mg/sqm; 125 mg/sqm or 150 mg/sqm)

SUMMARY:
An upfront-intensified treatment combining all the three active cytotoxic agents in metastatic colorectal cancer (mCRC) including fluoropyrimidines, oxaliplatin, irinotecan (FOLFOXIRI) plus antiangiogenic blockade with bevacizumab significantly improved survival. No biomarkers are available for predicting sensitivity/resistance to single chemotherapeutic drugs, the simultaneous delivery of all active chemotherapeutic agents might overcome resistance to single drugs.

Temozolomide has modest but non-negligible activity (about 10%) in chemo-refractory patients with MGMT methylated mCRC. The response rate to temozolomide-based therapy in pretreated patients is increased to up to 20% when restricting the focus on those with MGMT IHC-negative/MGMT methylated and MSS cancers. Clinical and preclinical synergy has been reported for combination of temozolomide with irinotecan and fluoropyrimidines. Temozolomide could be regarded as a "targeted" chemotherapy for patients with MSS and MGMT silenced tumors. In this subgroup of patients, an intensified triplet upfront regimen including temozolomide, fluoropyrimidines, irinotecan, associated with bevacizumab, could be a novel combination in molecularly super-selected mCRC patients.

Moving from this, the investigators designed this open-label, monocentric, phase 1b study evaluating the safety of the combination regimen 5-fluorouracil, leucovorin, irinotecan, temozolomide and bevacizumab in patients with MGMT silenced and MSS mCRC.

The study will consist in a dose-escalation assessment of the safety of the treatment in subjects with previously untreated MGMT silenced, MSS mCRC. A 3 + 3 design will be used to assess the maximum tolerated dose (MTD) or maximum tested dose of the combination FLIRT-bevacizumab. Upon completion of the phase 1b part, the phase 2 part of the study will start.

DETAILED DESCRIPTION:
An upfront-intensified treatment combining all the three active cytotoxic agents in mCRC including fluoropyrimidines, oxaliplatin, irinotecan (FOLFOXIRI) plus antiangiogenic blockade with bevacizumab significantly improved progression-free survival (PFS), overall survival (OS) and objective response rate (ORR) compared to standard FOLFIRI and bevacizumab irrespective to RAS/BRAF status, at price of higher rate of specific toxicities. Advantages of an intensified regimen include: 1) exposure to all active available drugs, since more than 10-15% of patients would not receive any second-line therapy due to early performance status deterioration; 2) the chance of achieving a high rate (around 36%) of secondary R0/R1 resection of metastases in patients with liver-limited and initially unresectable liver metastases.

Furthermore, results from the phase 3 TRIBE2 study showed that the intensified upfront regimen FOLFOXIRI-bevacizumab followed by the pre-planned reintroduction of the same agents after progressive disease provided a statistically significant and clinically relevant survival benefit when compared with the pre-planned sequential administration of FOLFOX-bevacizumab and FOLFIRI-bevacizumab in unresectable patients with mCRC. Therefore, FOLFOXIRI-bevacizumab regimen is recommended by all major guidelines as one of the possible upfront treatment options for mCRC, and is used in the clinical practice mainly for patients with highly aggressive disease (such as those with right sided and/or RAS or BRAF mutated). Notably, since no biomarkers are available for predicting sensitivity/resistance to single chemotherapeutic drugs, the simultaneous delivery of all active chemotherapeutic agents might overcome resistance to single drugs.

MGMT promoter methylation is found in about 40% of colorectal tumors. MGMT deficiency impairs DNA repair following administration of several alkylating agents, including temozolomide. Temozolomide has limited single-agent activity (around 10%) in patients with pretreated MGMT methylated mCRC. Promising activity has been reported for temozolomide in combination with the potentially synergic drug irinotecan (TEMIRI regimen) in clinically and molecularly selected patients. In a recent phase 2 randomized trial, capecitabine in combination with temozolomide (CAPTEM regimen) displayed similar activity and efficacy with respect to standard FOLFIRI as second-line therapy for MGMT methylated RAS mutated mCRC.

Heterogeneity of MGMT promoter methylation and residual MGMT protein expression might account for lack of activity of temozolomide in patients with MGMT promoter methylation assessed by means of a qualitative-only assay, i.e. methylation-specific PCR (MSP), which has been used as selection assay for patients' enrollment in published trials. Exploratory analyses have consistently shown the role of quantitative assessment of MGMT promoter methylation by means of digital PCR (methylBEAMing) and MGMT protein expression by immunohistochemistry (IHC) as potential predictive factors in mCRC patients treated with temozolomide. In the randomized phase 2 CAPTEM versus FOLFIRI second-line trial, patients with retained MGMT positivity by IHC had poorer outcomes in terms of PFS, OS and disease control rate (DCR: interaction test with arm: P=0.028). Any residual MGMT protein expression has been associated with lack of response to temozolomide across different trials, further supporting the restriction of temozolomide-based therapies for patients with MGMT IHC negativity coupled with gene methylation (MGMT silencing).

Mismatch repair deficiency/microsatellite instability (MSI) has been linked to innate resistance to several alkylating chemotherapeutic agents, including temozolomide, since cytotoxicity of these agents strictly relies on functional mismatch repair. Therefore, patients with MSI-high mCRC are excluded from temozolomide-based therapy.

Temozolomide could be regarded as a "targeted" chemotherapy for patients with MSS and MGMT silenced tumors. In this subgroup of patients, an intensified triplet upfront regimen including temozolomide, fluoropyrimidines, irinotecan, associated with bevacizumab, could be a novel combination in molecularly hyperselected mCRC patients.

Moving from this rationale the investigators designed this phase 1b trial assessing safety, recommended dose and preliminary activity of 5-fluoruracil, irinotecan, temozolomide and bevacizumab (FLIRT-bevacizumab) as a biomarker-guided initial therapy for patients with MGMT silenced and MSS mCRC.

The study will consist in a dose-escalation assessment of the safety of the treatment in subjects with previously untreated MGMT silenced, MSS mCRC.

A 3 + 3 design will be used to assess the maximum tolerated dose (MTD) or maximum tested dose of the combination FLIRT-bevacizumab.

The MTD will be defined as the dose level at which ≥2/3 or ≥2/6 subjects experience a dose-limiting toxicity (DLT). When the MTD or maximum tested dose has been determined or reached, the RP2D to be tested in a future phase II trial will be one dose level below the MTD or the maximum tested dose if MTD will not be reached. At least 6 patients should be treated at the RD during the dose escalation.

The treatment will consist of an induction period of four 28-day cycles of FLIRT- bevacizumab followed by maintenance regimen of 5-FU/LV-bevacizumab administered every 14 days in combination with per os temozolomide according to dose level over days 1-5 every 28 days in patients without progressive disease at the end of the induction period. Patients will undergo tumor assessment at baseline and every 8 ± 1 weeks until confirmed disease progression, unacceptable toxicity, withdrawal of consent, death, whichever occurs first. The treatment will continue until progressive disease, unacceptable toxicities, or consent withdrawal.

The phase 1b part of the study has been completed and the RP2D of temozolomide is 150 mg/sqm on days 1-5 every 28 days. The phase 2 part is ongoing.

ELIGIBILITY:
(applies to phase 2 part)

Inclusion criteria

1. Histologically confirmed metastatic adenocarcinoma of the colon and/or rectum.
2. Confirmed MGMT promoter methylation by PSQ (> 5%) and absent MGMT expression by immunohistochemistry.
3. Locally assessed pMMR or MSS status.
4. Written informed consent obtained prior to any study procedures.
5. Availability of archival tumor tissue (primary tumor and metastases or at least one of the two) for confirmation of MGMT, MMR/MSI status and biomarker analyses.
6. Availability of blood sample for biomarker analysis.
7. Metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
8. At least one measurable lesion according to RECIST 1.1.
9. Age ≥ 18 and less or equal than 75 years.
10. ECOG PS ≤ 1 if patient < 70 years old; ECOG PS 0 if patient 70-75 years old.
11. Life expectancy of at least 12 weeks.
12. Previous (neo)adjuvant fluoropyrimidine or fluoropyrimidine plus oxaliplatin chemotherapy allowed only if more than 6 months elapsed between the end of (neo)adjuvant therapy and first evidence of disease relapse.
13. Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hemoglobin ≥ 9 g/dl.
14. Total bilirubin ≤1.5 fold the upper-normal limits (UNL), AST (SGOT) and/or ALT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases).
15. Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL.
16. Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of amenorrhea, a single FSH measurement is insufficient.
17. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must be willing to use adequate contraception as approved be the Investigator (barrier contraceptive measure or oral contraception) as outlined in Section 7.6, starting with the screening visit and through 6 months after the last treatment dose. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
18. Will and ability to comply with the protocol.
19. Is willing and able to provide an adequate archival tumor sample (FFPE) available for molecular screening and exploratory analyses. If the tumor block is not available, a minimum of 25 3-micron unstained sections on charged slides of tumor will be required.

Exclusion criteria

1. Requirement for treatment with any medicinal product that contraindicates the use of any of the study medications, may interfere with the planned treatment, affects patient compliance or puts the patient at high risk for treatment-related complications.
2. Metastatic disease deemed R0 resectable upfront or after induction therapy by means of multidisciplinary team assessment.
3. Radiotherapy to any site within 4 weeks before the study.
4. Presence of one of the following: DPYD2a (c.1905+1G>A); DPYD13 (c.1679 T>G); DPYD D949V (c.2846 A>T); DPYD IVS10 (c.1129-5923 C>G).
5. Presence of one of the following UGT1A1 1(TA)6/UGT1A1 36(TA)5; UGT1A1 28(TA)7/UGT1A1 37(TA)8 (homozygous genotype).
6. In the dose escalation phase, untreated brain metastases or spinal cord compression or primary brain tumors; in the dose expansion phase, known history of brain metastases.
7. History or evidence upon physical examination of central nervous system disease unless adequately treated.8. Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration.

9. Evidence of bleeding diathesis or coagulopathy. 10. Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.

11. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.

12. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.

13. Any previous venous thromboembolism ≥ NCI CTCAE Grade 4. 14. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to the first study treatment.

15. Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer).

16. Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.

17. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.

18. Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.

19. Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.

20. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
(Phase 1b) safety and to determine the recommended phase 2 dose of the combination of FLIRT- bevacizumab in patients with MGMT silenced and MSS mCRC, previously untreated for advanced disease. (Phase 2) efficacy of FLIRT/bev | 24 months
  (phase 1b) The RD to be tested in a future phase 2 trial will be one dose level below the MTD or the maximum tested dose if MTD will not be reached. he MTD will be defined as the dose level at which ≥2/3 or ≥2/6 subjects experience a dose-limiting toxicity. At least 6 patients should be treated at the RD during the dose escalation.
  (phase 2) an overall sample size of 27 patients achieves an 80% power to detect the probability to increase 9-month PFS rate to 55% with a one-sided α level of 0.1 by the combination of temozolomide at the RP2D in combination with irinotecan, 5-fluorouracil and bevacizumab. The null hypothesis will be rejected if at least 14 patients are free of disease progression at 9 months.

SECONDARY OUTCOMES:
ORR obtained by FLIRT bevacizumab | 24 months
  To assess ORR per RECIST version 1.1
Quality of life as assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 24 months
  EORTC QLQ-C30 administered every 8 weeks
Quality of life as assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29) | 24 months
  EORTC QLQ-CR29 administered every 8 weeks
Quality of life as assessed using the Euro Quality of Life 5 Dimensions Questionnaire (EQ-5D-5L) | 24 months
  EQ-5D-5L administered every 8 weeks

OTHER OUTCOMES:
OS of FLIRT bevacizumab (phase 2) - secondary endpoint for phase 2 | 24 months
  OS is defined as the time from enrolment to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Evaluate tumor biomarkers in archival tumor tissue | 24 months
  Quantification of the percentage of MGMT methylation by digital PCR methylBEAMing will be performed in archival tumor tissue. Mutational load will be assessed in archival tumor tissues by means of whole exome sequencing.
Evaluate plasma biomarkers in longitudinal blood samples (plasma and PBMCs) | 24 months
  Digital PCR for MGMT methylation status will be performed in cell-free circulating DNA (cfDNA). Mutational load will be assessed in cfDNA by means of whole exome sequencing.
PFS of FLIRT bevacizumab (phase 1b) | 24 months
  FS is defined as the time from enrolment to the first documentation of objective disease progression determined by investigator assessment or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumour assessment documenting absence of progressive disease for patients who are alive, on study and progression free at the time of the analysis. Alive patients having no tumour assessments after baseline will have time to event censored on the date of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (3):
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan
  - Istituto Oncologico Veneto IRCCS, Padua, PD
  - Ospedale Santa Chiara, Pisa, PI

REFERENCES:
- [Background] Yoshino T, Arnold D, Taniguchi H, Pentheroudakis G, Yamazaki K, Xu RH, Kim TW, Ismail F, Tan IB, Yeh KH, Grothey A, Zhang S, Ahn JB, Mastura MY, Chong D, Chen LT, Kopetz S, Eguchi-Nakajima T, Ebi H, Ohtsu A, Cervantes A, Muro K, Tabernero J, Minami H, Ciardiello F, Douillard JY. Pan-Asian adapted ESMO consensus guidelines for the management of patients with metastatic colorectal cancer: a JSMO-ESMO initiative endorsed by CSCO, KACO, MOS, SSO and TOS. Ann Oncol. 2018 Jan 1;29(1):44-70. doi: 10.1093/annonc/mdx738. PMID 29155929
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126
- [Background] Douillard JY, Cunningham D, Roth AD, Navarro M, James RD, Karasek P, Jandik P, Iveson T, Carmichael J, Alakl M, Gruia G, Awad L, Rougier P. Irinotecan combined with fluorouracil compared with fluorouracil alone as first-line treatment for metastatic colorectal cancer: a multicentre randomised trial. Lancet. 2000 Mar 25;355(9209):1041-7. doi: 10.1016/s0140-6736(00)02034-1. PMID 10744089
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366
- [Background] Sorich MJ, Wiese MD, Rowland A, Kichenadasse G, McKinnon RA, Karapetis CS. Extended RAS mutations and anti-EGFR monoclonal antibody survival benefit in metastatic colorectal cancer: a meta-analysis of randomized, controlled trials. Ann Oncol. 2015 Jan;26(1):13-21. doi: 10.1093/annonc/mdu378. Epub 2014 Aug 12. PMID 25115304
- [Background] Holch JW, Ricard I, Stintzing S, Modest DP, Heinemann V. The relevance of primary tumour location in patients with metastatic colorectal cancer: A meta-analysis of first-line clinical trials. Eur J Cancer. 2017 Jan;70:87-98. doi: 10.1016/j.ejca.2016.10.007. Epub 2016 Nov 29. PMID 27907852
- [Background] Falcone A, Masi G, Allegrini G, Danesi R, Pfanner E, Brunetti IM, Di Paolo A, Cupini S, Del Tacca M, Conte P. Biweekly chemotherapy with oxaliplatin, irinotecan, infusional Fluorouracil, and leucovorin: a pilot study in patients with metastatic colorectal cancer. J Clin Oncol. 2002 Oct 1;20(19):4006-14. doi: 10.1200/JCO.2002.12.075. PMID 12351598
- [Background] Masi G, Allegrini G, Cupini S, Marcucci L, Cerri E, Brunetti I, Fontana E, Ricci S, Andreuccetti M, Falcone A. First-line treatment of metastatic colorectal cancer with irinotecan, oxaliplatin and 5-fluorouracil/leucovorin (FOLFOXIRI): results of a phase II study with a simplified biweekly schedule. Ann Oncol. 2004 Dec;15(12):1766-72. doi: 10.1093/annonc/mdh470. PMID 15550581
- [Background] Masi G, Loupakis F, Salvatore L, Fornaro L, Cremolini C, Cupini S, Ciarlo A, Del Monte F, Cortesi E, Amoroso D, Granetto C, Fontanini G, Sensi E, Lupi C, Andreuccetti M, Falcone A. Bevacizumab with FOLFOXIRI (irinotecan, oxaliplatin, fluorouracil, and folinate) as first-line treatment for metastatic colorectal cancer: a phase 2 trial. Lancet Oncol. 2010 Sep;11(9):845-52. doi: 10.1016/S1470-2045(10)70175-3. Epub 2010 Aug 9. PMID 20702138
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Grothey A, Sargent D, Goldberg RM, Schmoll HJ. Survival of patients with advanced colorectal cancer improves with the availability of fluorouracil-leucovorin, irinotecan, and oxaliplatin in the course of treatment. J Clin Oncol. 2004 Apr 1;22(7):1209-14. doi: 10.1200/JCO.2004.11.037. PMID 15051767
- [Background] Cremolini C, Casagrande M, Loupakis F, Aprile G, Bergamo F, Masi G, Moretto R R, Pietrantonio F, Marmorino F, Zucchelli G, Tomasello G, Tonini G, Allegrini G, Granetto C, Ferrari L, Urbani L, Cillo U, Pilati P, Sensi E, Pellegrinelli A, Milione M, Fontanini G, Falcone A. Efficacy of FOLFOXIRI plus bevacizumab in liver-limited metastatic colorectal cancer: A pooled analysis of clinical studies by Gruppo Oncologico del Nord Ovest. Eur J Cancer. 2017 Mar;73:74-84. doi: 10.1016/j.ejca.2016.10.028. Epub 2016 Dec 13. PMID 27986363
- [Background] Pietrantonio F, Cotsoglou C, Fuca G, Lo Vullo S, Nichetti F, Milione M, Coppa J, Vaiani M, Alessi A, Prisciandaro M, Droz-Dit Busset M, Morano F, Corallo S, Lazzati S, Antista M, Mennitto A, Randon G, Raimondi A, Belfiore A, Padovano B, Perrone F, Mariani L, Di Bartolomeo M, de Braud F, Mazzaferro V. Perioperative Bevacizumab-based Triplet Chemotherapy in Patients With Potentially Resectable Colorectal Cancer Liver Metastases. Clin Colorectal Cancer. 2019 Mar;18(1):34-43.e6. doi: 10.1016/j.clcc.2018.11.004. Epub 2018 Nov 24. PMID 30558859
- [Background] Cremolini C, Antoniotti C, Rossini D, Lonardi S, Loupakis F, Pietrantonio F, Bordonaro R, Latiano TP, Tamburini E, Santini D, Passardi A, Marmorino F, Grande R, Aprile G, Zaniboni A, Murgioni S, Granetto C, Buonadonna A, Moretto R, Corallo S, Cordio S, Antonuzzo L, Tomasello G, Masi G, Ronzoni M, Di Donato S, Carlomagno C, Clavarezza M, Ritorto G, Mambrini A, Roselli M, Cupini S, Mammoliti S, Fenocchio E, Corgna E, Zagonel V, Fontanini G, Ugolini C, Boni L, Falcone A; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab and reintroduction after progression versus mFOLFOX6 plus bevacizumab followed by FOLFIRI plus bevacizumab in the treatment of patients with metastatic colorectal cancer (TRIBE2): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2020 Apr;21(4):497-507. doi: 10.1016/S1470-2045(19)30862-9. Epub 2020 Mar 9. PMID 32164906
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Fu D, Calvo JA, Samson LD. Balancing repair and tolerance of DNA damage caused by alkylating agents. Nat Rev Cancer. 2012 Jan 12;12(2):104-20. doi: 10.1038/nrc3185. PMID 22237395
- [Background] Esteller M, Herman JG. Generating mutations but providing chemosensitivity: the role of O6-methylguanine DNA methyltransferase in human cancer. Oncogene. 2004 Jan 8;23(1):1-8. doi: 10.1038/sj.onc.1207316. PMID 14712205
- [Background] Hochhauser D, Glynne-Jones R, Potter V, Gravalos C, Doyle TJ, Pathiraja K, Zhang Q, Zhang L, Sausville EA. A phase II study of temozolomide in patients with advanced aerodigestive tract and colorectal cancers and methylation of the O6-methylguanine-DNA methyltransferase promoter. Mol Cancer Ther. 2013 May;12(5):809-18. doi: 10.1158/1535-7163.MCT-12-0710. Epub 2013 Feb 26. PMID 23443801
- [Background] Pietrantonio F, Perrone F, de Braud F, Castano A, Maggi C, Bossi I, Gevorgyan A, Biondani P, Pacifici M, Busico A, Gariboldi M, Festinese F, Tamborini E, Di Bartolomeo M. Activity of temozolomide in patients with advanced chemorefractory colorectal cancer and MGMT promoter methylation. Ann Oncol. 2014 Feb;25(2):404-8. doi: 10.1093/annonc/mdt547. Epub 2013 Dec 29. PMID 24379162
- [Background] Pietrantonio F, de Braud F, Milione M, Maggi C, Iacovelli R, Dotti KF, Perrone F, Tamborini E, Caporale M, Berenato R, Leone G, Pellegrinelli A, Bossi I, Festinese F, Federici S, Di Bartolomeo M. Dose-Dense Temozolomide in Patients with MGMT-Silenced Chemorefractory Colorectal Cancer. Target Oncol. 2016 Jun;11(3):337-43. doi: 10.1007/s11523-015-0397-2. PMID 26538496
- [Background] Amatu A, Barault L, Moutinho C, Cassingena A, Bencardino K, Ghezzi S, Palmeri L, Bonazzina E, Tosi F, Ricotta R, Cipani T, Crivori P, Gatto R, Chirico G, Marrapese G, Truini M, Bardelli A, Esteller M, Di Nicolantonio F, Sartore-Bianchi A, Siena S. Tumor MGMT promoter hypermethylation changes over time limit temozolomide efficacy in a phase II trial for metastatic colorectal cancer. Ann Oncol. 2016 Jun;27(6):1062-1067. doi: 10.1093/annonc/mdw071. Epub 2016 Feb 24. PMID 26916096
- [Background] Calegari MA, Inno A, Monterisi S, Orlandi A, Santini D, Basso M, Cassano A, Martini M, Cenci T, de Pascalis I, Camarda F, Barbaro B, Larocca LM, Gori S, Tonini G, Barone C. A phase 2 study of temozolomide in pretreated metastatic colorectal cancer with MGMT promoter methylation. Br J Cancer. 2017 May 9;116(10):1279-1286. doi: 10.1038/bjc.2017.109. Epub 2017 Apr 20. PMID 28427088
- [Background] Sartore-Bianchi A, Pietrantonio F, Amatu A, Milione M, Cassingena A, Ghezzi S, Caporale M, Berenato R, Falcomata C, Pellegrinelli A, Bardelli A, Nichelatti M, Tosi F, De Braud F, Di Nicolantonio F, Barault L, Siena S. Digital PCR assessment of MGMT promoter methylation coupled with reduced protein expression optimises prediction of response to alkylating agents in metastatic colorectal cancer patients. Eur J Cancer. 2017 Jan;71:43-50. doi: 10.1016/j.ejca.2016.10.032. Epub 2016 Dec 18. PMID 27997874
- [Background] Pietrantonio F, Lobefaro R, Antista M, Lonardi S, Raimondi A, Morano F, Mosconi S, Rimassa L, Murgioni S, Sartore-Bianchi A, Tomasello G, Longarini R, Farina G, Petrelli F, Gori S, Randon G, Corallo S, Pagani F, Guarini V, Palermo F, Martinetti A, Macagno M, Barault L, Perrone F, Tamborini E, Milione M, Di Nicolantonio F, Di Maio M, Fuca G, Di Bartolomeo M, de Braud F. Capecitabine and Temozolomide versus FOLFIRI in RAS-Mutated, MGMT-Methylated Metastatic Colorectal Cancer. Clin Cancer Res. 2020 Mar 1;26(5):1017-1024. doi: 10.1158/1078-0432.CCR-19-3024. Epub 2019 Nov 18. PMID 31740551
- [Background] Morano F, Corallo S, Niger M, Barault L, Milione M, Berenato R, Moretto R, Randon G, Antista M, Belfiore A, Raimondi A, Nichetti F, Martinetti A, Battaglia L, Perrone F, Pruneri G, Falcone A, Di Bartolomeo M, de Braud F, Di Nicolantonio F, Cremolini C, Pietrantonio F. Temozolomide and irinotecan (TEMIRI regimen) as salvage treatment of irinotecan-sensitive advanced colorectal cancer patients bearing MGMT methylation. Ann Oncol. 2018 Aug 1;29(8):1800-1806. doi: 10.1093/annonc/mdy197. PMID 29860358
- [Background] Pietrantonio F, Randon G, Romagnoli D, Di Donato S, Benelli M, de Braud F. Biomarker-guided implementation of the old drug temozolomide as a novel treatment option for patients with metastatic colorectal cancer. Cancer Treat Rev. 2020 Jan;82:101935. doi: 10.1016/j.ctrv.2019.101935. Epub 2019 Nov 28. PMID 31821983
- [Background] Fine RL, Gulati AP, Krantz BA, Moss RA, Schreibman S, Tsushima DA, Mowatt KB, Dinnen RD, Mao Y, Stevens PD, Schrope B, Allendorf J, Lee JA, Sherman WH, Chabot JA. Capecitabine and temozolomide (CAPTEM) for metastatic, well-differentiated neuroendocrine cancers: The Pancreas Center at Columbia University experience. Cancer Chemother Pharmacol. 2013 Mar;71(3):663-70. doi: 10.1007/s00280-012-2055-z. Epub 2013 Jan 31. PMID 23370660
- [Background] Houghton PJ, Stewart CF, Cheshire PJ, Richmond LB, Kirstein MN, Poquette CA, Tan M, Friedman HS, Brent TP. Antitumor activity of temozolomide combined with irinotecan is partly independent of O6-methylguanine-DNA methyltransferase and mismatch repair phenotypes in xenograft models. Clin Cancer Res. 2000 Oct;6(10):4110-8. PMID 11051264
- [Background] Pourquier P, Waltman JL, Urasaki Y, Loktionova NA, Pegg AE, Nitiss JL, Pommier Y. Topoisomerase I-mediated cytotoxicity of N-methyl-N'-nitro-N-nitrosoguanidine: trapping of topoisomerase I by the O6-methylguanine. Cancer Res. 2001 Jan 1;61(1):53-8. PMID 11196197
- [Background] Newlands ES, Blackledge GR, Slack JA, Rustin GJ, Smith DB, Stuart NS, Quarterman CP, Hoffman R, Stevens MF, Brampton MH, et al. Phase I trial of temozolomide (CCRG 81045: M&B 39831: NSC 362856). Br J Cancer. 1992 Feb;65(2):287-91. doi: 10.1038/bjc.1992.57. PMID 1739631
- [Background] Pitot HC, Goldberg RM, Reid JM, Sloan JA, Skaff PA, Erlichman C, Rubin J, Burch PA, Adjei AA, Alberts SA, Schaaf LJ, Elfring G, Miller LL. Phase I dose-finding and pharmacokinetic trial of irinotecan hydrochloride (CPT-11) using a once-every-three-week dosing schedule for patients with advanced solid tumor malignancy. Clin Cancer Res. 2000 Jun;6(6):2236-44. PMID 10873073
- [Background] Sobrero AF, Aschele C, Bertino JR. Fluorouracil in colorectal cancer--a tale of two drugs: implications for biochemical modulation. J Clin Oncol. 1997 Jan;15(1):368-81. doi: 10.1200/JCO.1997.15.1.368. PMID 8996164
- [Background] Bardelli A, Cahill DP, Lederer G, Speicher MR, Kinzler KW, Vogelstein B, Lengauer C. Carcinogen-specific induction of genetic instability. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5770-5. doi: 10.1073/pnas.081082898. Epub 2001 Apr 10. PMID 11296254
- [Background] Cahill DP, Levine KK, Betensky RA, Codd PJ, Romany CA, Reavie LB, Batchelor TT, Futreal PA, Stratton MR, Curry WT, Iafrate AJ, Louis DN. Loss of the mismatch repair protein MSH6 in human glioblastomas is associated with tumor progression during temozolomide treatment. Clin Cancer Res. 2007 Apr 1;13(7):2038-45. doi: 10.1158/1078-0432.CCR-06-2149. PMID 17404084
- [Background] Alexandrov LB, Stratton MR. Mutational signatures: the patterns of somatic mutations hidden in cancer genomes. Curr Opin Genet Dev. 2014 Feb;24(100):52-60. doi: 10.1016/j.gde.2013.11.014. Epub 2013 Dec 29. PMID 24657537
- [Background] Coffield VM, Helms WS, Jiang Q, Su L. Galpha13 mediates a signal that is essential for proliferation and survival of thymocyte progenitors. J Exp Med. 2004 Nov 15;200(10):1315-24. doi: 10.1084/jem.20040944. Epub 2004 Nov 8. PMID 15534370
- [Background] Hervieu A, Rebe C, Vegran F, Chalmin F, Bruchard M, Vabres P, Apetoh L, Ghiringhelli F, Mignot G. Dacarbazine-mediated upregulation of NKG2D ligands on tumor cells activates NK and CD8 T cells and restrains melanoma growth. J Invest Dermatol. 2013 Feb;133(2):499-508. doi: 10.1038/jid.2012.273. Epub 2012 Sep 6. PMID 22951720
- [Background] Germano G, Lamba S, Rospo G, Barault L, Magri A, Maione F, Russo M, Crisafulli G, Bartolini A, Lerda G, Siravegna G, Mussolin B, Frapolli R, Montone M, Morano F, de Braud F, Amirouchene-Angelozzi N, Marsoni S, D'Incalci M, Orlandi A, Giraudo E, Sartore-Bianchi A, Siena S, Pietrantonio F, Di Nicolantonio F, Bardelli A. Inactivation of DNA repair triggers neoantigen generation and impairs tumour growth. Nature. 2017 Dec 7;552(7683):116-120. doi: 10.1038/nature24673. Epub 2017 Nov 29. PMID 29186113
- [Background] Lu Y, Zhao Z, Wang J, Lv W, Lu L, Fu W, Li W. Safety and efficacy of combining capecitabine and temozolomide (CAPTEM) to treat advanced neuroendocrine neoplasms: A meta-analysis. Medicine (Baltimore). 2018 Oct;97(41):e12784. doi: 10.1097/MD.0000000000012784. PMID 30313101